CLINICAL TRIAL: NCT05661968
Title: Efficacy of an Online Educational Program to Change Back Pain Beliefs in Physical Therapists: a Randomized Controlled Trial
Brief Title: Efficacy of an Online Educational Program to Change Back Pain Beliefs in Physical Therapists
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Rafael Zambelli Pinto, Lecturer, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAAE 60756422.6.0000.5149
Record Dates: First submitted 2022-12-14; First posted 2022-12-22 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Low Back Pain
Keywords: Low back pain; Online educational program; Beliefs; Physical Therapists
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online educational program (Experimental): A 6-week educational program delivered online based on information and recommendations from international clinical practice guidelines for the management of back pain.
  Interventions: Other: Online educational program
- Control group (No Intervention): The control group will receive no intervention and will be instructed to follow their clinical practice normally.

INTERVENTIONS:
Other: Online educational program — The intervention group will receive an online educational program, containing current information on low back pain management according to international clinical practice guidelines. Program content includes recommendations on assessment, diagnosis, and treatment of low back pain. The online program has 6 units of studies, with the content offered in the formats of video classes, infographics, texts, websites and clinical cases. The participant must complete the course within 6 weeks and will be able to set their own pace. Participants in the intervention group will receive their login and access password via email.
  Arms: Online educational program

SUMMARY:
The goal of this clinical trial is to investigate the efficacy of an online educational program for physical therapists to change back pain beliefs. The main questions it aims to answer are:

- What is the effect of an online educational program to change beliefs about the management of back pain in physical therapists?

A total of 106 physical therapists will be recruited for this study. Participants will be randomized into two groups: intervention and control groups. The intervention group will receive a 6-week online educational program including recommendations from international clinical practice guidelines for the management of back pain. The control group will not receive any intervention. The outcomes of this trial include beliefs about management of back pain and imaging exams and will be assessed at baseline and 6 weeks after randomization.

ELIGIBILITY:
Inclusion Criteria:

* must be a licensed physical therapist;
* currently managing patients with low back pain, regardless of the duration of symptoms, in clinical practice;
* if not currently managing patients with low back pain, participants must have treated at least one patient in the last month.

(Patients with low back pain are defined as those patients reporting pain between the lower border of the last vertebral ribs and the gluteal fold, with or without pain referred to the lower limb).

Exclusion Criteria:

* not having access or reporting difficulty in accessing the internet.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-07-28 (Actual); Study Completion 2023-07-28 (Actual)

PRIMARY OUTCOMES:
Modified Back Belief Questionnaire | Post-intervention (i.e. 6 weeks after randomization)
  This questionnaire consists of 25 items assessing the following aspects: low back pain outcomes at work and patients' social life, treatment (including medication, surgical procedures, alternative treatments), low back pain prognosis, causes of low back pain and diagnostic methods. The score of each item follows a Likert scale ranging from 1 to 5, where each items mean, 1. "Completely Disagree"; 2. Disagree; 3. "I neither agree nor disagree"; 4. "Agree" and 5; "Completely Agree". To calculate the final score of the questionnaire, the score of each item on the Likert scale is transformed into a score ranging from -2 to 2. The total score of the questionnaire ranges from -50 to 50 points, with values closest to 50 points indicate more adequate beliefs regarding low back pain.

SECONDARY OUTCOMES:
Back Pain Attitudes Questionnaire (Back-PAQ) | Post-intervention (i.e. 6 weeks after randomization)
  The items in this questionnaire comprise general aspects related to low back pain, including beliefs about pain-related behavior and symptom recovery. The short version of the questionnaire with 10 items will be used. Each item is scored on a 5-point Likert scale. The total score of the questionnaire ranges from -20 to 20, with lower values (or closer to 20) indicating more adequate beliefs.
Beliefs regarding imaging exams | Post-intervention (i.e. 6 weeks after randomization)
  Beliefs regarding imaging exams will be measured using two statements from a previous study5: Q1- 'X-rays or scans are necessary to get the best medical care for low back pain'; Q2 - 'Everyone with low back pain should have spine imaging (e.g. X-ray, computed tomography or magnetic resonance imaging)'. Participants indicated their agreement with each statement on a 5-point Likert scale of 'Strongly Disagree' (1) to 'Strongly Agree' (5). The 5-point Likert responses will be dichotomised into two categories: correct beliefs (disagree or strongly disagree) and incorrect beliefs (neither agree nor disagree, agree or strongly agree) about imaging prescription.

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Z Pinto, PhD, Principal Investigator — Universidade Federal de Minas Geral
Locations (1):
- Universidade Federal de Minas Gerais, Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Diniz LM, Oliveira CB, Machado GC, Maher CG, Verhagen AP, Fernandes DAM, Franco MR, Souza TR, Pinto RZ. Effectiveness of brief patient information materials for promoting correct beliefs about imaging and inevitable consequences of low back pain: A randomised controlled trial. Clin Rehabil. 2022 Apr;36(4):527-537. doi: 10.1177/02692155211065974. Epub 2021 Dec 21. PMID 34931854
- [Background] Fernandes DAM, Freire APCF, Santos JM, Lemes IR, Diniz LM, FRANCO, MR, Ocarino JM, Pinto RZ. The Modified Back Beliefs Questionnaire as a tool to screen for incorrect beliefs regarding back pain: Cross-cultural adaptation and measurement properties. International Journal of Osteopathic Medicine. 2022; 44: 9-15. https://doi.org/10.1016/j.ijosm.2022.04.001
- [Derived] Magalhaes DS, McAuley JH, Maher CG, Ferreira EMR, Oliveira TEP, Mastahinich MER, de Jesus-Moraleida FR, Fukusawa L, Franco MR, Pinto RZ. An e-learning program improves low back pain beliefs of physiotherapists: a randomised trial. J Physiother. 2025 Jan;71(1):35-41. doi: 10.1016/j.jphys.2024.11.014. Epub 2024 Dec 14. PMID 39675949